CLINICAL TRIAL: NCT07167550
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Comparative Study of the Efficacy and Safety of the Drug Dimephosphon®, Concentrate for Solution for Intravenous Administration, 1 g, in Acute Ischemic Stroke Patients
Brief Title: The Study of Efficacy and Safety of Dimephosphon® in Acute Ischemic Stroke
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tatchempharmpreparaty, JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMF-III-24; DMF-III-24 (Other: Tatchempharmpreparaty, JSC)
Record Dates: First submitted 2025-09-03; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Acute Stroke; Ischemic Stroke; Cerebrovascular Disorders; Physiological Effects of Drugs
Keywords: Neuroprotective Agents; Protective Agents; Neuroprotection; Anti-acidemic agents; Dimephosphon; Dimethyloxobutylphosphonyldimethylate; Acute Stroke; Ischemic Stroke; Antioxidants
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebrovascular Disorders | interventions — dimephosphon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dimephosphon® (Experimental): Days 1-3: Dimephosphon® 2 g (2 vials) administered as intravenous infusion diluted in 200 mL of 0.9% sodium chloride solution three times daily (morning, afternoon, and evening, with minimum 5-hour interval between administrations).
  Days 4-14: Dimephosphon® 2 g (2 vials) administered as intravenous bolus diluted in 20 mL of 0.9% sodium chloride solution three times daily (morning, afternoon, and evening, with minimum 5-hour interval between administrations).
  Interventions: Drug: Dimephosphon®
- Placebo (Placebo Comparator): Days 1-3: Placebo 2 g (2 vials) administered as intravenous infusion diluted in 200 mL of 0.9% sodium chloride solution three times daily (morning, afternoon, and evening, with minimum 5-hour interval between administrations).
  Days 4-14: Placebo 2 g (2 vials) administered as intravenous bolus diluted in 20 mL of 0.9% sodium chloride solution three times daily (morning, afternoon, and evening, with minimum 5-hour interval between administrations).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimephosphon® — 1 g/ml, concentrate for solution for intravenous infusion
  Arms: Dimephosphon®
Drug: Placebo — Placebo IV solution
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of Dimephosphon® in acute ischemic stroke

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled trial. The purpose of the study is to evaluate the efficacy and safety of Dimephosphon® in acute ischemic stroke. The study includes a screening period (Visit 1, up to 48 hours) and a treatment period (Visits 2-4). Subjects will be randomized into 2 groups in a 1:1 ratio: Group A (investigational drug Dimephosphon®) and Group B (placebo). Key inclusion criteria: verified by CT/MRI current hemispheric ischemic stroke, NIHSS score ≥5 and ≤15 at screening. The study will assess clinical outcomes using standardized scales including NIHSS, mRS, MMSE, MoCA and EQ-5D.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent was obtained from the patient or their legally authorized representative prior to study participation.
2. Age 35-80.
3. Patients must exhibit neurological manifestations consistent with acute ischemic stroke, with a documented onset-to-intervention interval ranging from 24 to 72 hours at the time of scheduled initial administration of the investigational drug.
4. Verified by CT/MRI current hemispheric ischemic stroke.
5. NIHSS score ≥5 and ≤15 at screening.
6. Ability to comply with all protocol-specified procedures, prohibitions, and restrictions.
7. Willingness and ability to adhere to highly effective contraceptive methods as outlined in the study protocol.

Exclusion Criteria:

1. Hemorrhagic stroke or hemorrhagic transformation of ischemic focus, traumatic brain injuries
2. Vertebrobasilar stroke and/or development of acute insufficiency syndromes in the arteries of the vertebrobasilar system
3. A patient with ischemic stroke who is a candidate for reperfusion therapy or who has undergone reperfusion therapy before participation in this study.
4. The presence of anatomical abnormalities of the cerebral vessels (arteriovenous malformations, cavernous malformations, aneurysms, atresia of at least one of the extracranial arteries) according to the anamnesis or CT/MRI data.
5. Progression of neurological symptoms of stroke, defined as an increase in the NIHSS score by 4 points at the second assessment (immediately before randomization) from the value obtained at the first assessment (immediately after signing the informed consent form).
6. Surgery on the carotid arteries less than 1 year before screening.
7. History of stroke less than 1 year before screening.
8. Myocardial infarction less than 6 months before screening.
9. Chronic renal failure stage 2-3 (creatinine clearance less than 40 ml/min).
10. Pregnancy or lactation.
11. Participation in another trial within 28 days prior to enrollment.
12. Use of prohibited medications.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-09-06 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects having Modified Rankin Scale (mRS) scores 0-2 at Visit 4 (Day 15) | Day 15

SECONDARY OUTCOMES:
Percentage of subjects having Modified Rankin Scale (mRS) scores 0-2 at Visit 3 (Day 8), Visit 5 (Day 30), Visit 6 (Day 90). | Day 8, Day 30, Day 90
Change from Baseline (Visit 1, no more than 48 hours) in the National Institutes of Health Stroke Scale (NIHSS) score at Visit 3 (Day 8), Visit 4 (Day 15), Visit 5 (Day 30), Visit 6 (Day 90). | Baseline, Day 8, Visit 4 Day 15, Day 30, Day 90
Percentage of subjects with changes from Baseline (Visit 1, no more than 48 hours) in NIHSS score at Visit 3 (Day 8), Visit 4 (Day 15), Visit 5 (Day 30), Visit 6 (Day 90). | Baseline, Day 8, Day 15, Day 30, Day 90
Proportion of patients with a ≥4-point change in NIHSS score from Baseline (Visit 1, no more than 48 hours) at Visit 3 (Day 8), Visit 4 (Day 15), Visit 5 (Day 30), and Visit 6 (Day 90). | Baseline, Day 8, Day 15, Day 30, Day 90
Proportion of patients with a ≥2-point change in NIHSS score from Baseline (Visit 1, no more than 48 hours) to Visit 3 (Day 8), Visit 4 (Day 15), Visit 5 (Day 30), Visit 6 (Day 90). | Baseline, Day 8, Day 15, Day 30, Day 90
Change from Baseline (Visit 1, no more than 48 hours) in the Montreal Cognitive Assessment (MoCA) score at Visit 3 (Day 8), Visit 4 (Day 15), Visit 5 (Day 30), Visit 6 (Day 90). | Baseline, Day 8, Day 15, Day 30, Day 90
Change from Baseline (Visit 1, no more than 48 hours) in the Mini-Mental State Examination (MMSE) score at Visit 3 (Day 8), Visit 4 (Day 15), Visit 5 (Day 30), Visit 6 (Day 90). | Baseline, Day 8, Day 15, Day 30, Day 90
Change from Baseline (Visit 1, no more than 48 hours) in the EuroQol 5-Dimensions (EQ-5D) score at Visit 3 (Day 8), Visit 4 (Day 15), Visit 5 (Day 30), Visit 6 (Day 90). | Baseline, Day 8, Day 15, Day 30, Day 90
All-cause mortality from Visit 2 to Visit 6 (Hazard Ratio) | up to Day 90

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - State Budgetary Healthcare Institution of the Leningrad Region "Vsevolozhsk Interdistrict Clinical Hospital, Vsevolozhsk, Leningradskaya Oblast'
  - State Budgetary Healthcare Institution "Research Institute - Regional Clinical Hospital No. 1 named after Professor S.V. Ochapovsky" of the Ministry of Health of the Krasnodar region, Krasnodar
  - Federal State Autonomous Educational Institution of Higher Education "Peoples' Friendship University of Russia named after Patrice Lumumba", Moscow
  - The FSBI "Federal Center of Brain Research and Neurotechnologies" of the Federal Medical and Biological Agency, Moscow
  - Saint Petersburg State Budgetary Healthcare Institution "City Hospital No. 40 of the Kurortny District", Saint Petersburg
  - State Budgetary Healthcare Institution "City Hospital No. 4 of Sochi" of the Ministry of Healthcare of the Krasnodar Region, Sochi